CLINICAL TRIAL: NCT06620419
Title: Clinical Evaluation of Perineal Electrical Stimulation for Urinary Incontinence in Men
Brief Title: Clinical Study of External Electrical Stimulation for Male Incontinence
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elidah, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR-1168
Record Dates: First submitted 2024-05-16; First posted 2024-10-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-10

CONDITIONS: Urinary Incontinence
Keywords: male; men; prostatetectomy; incontinence; electrical stimulation
MeSH Terms: conditions — Urinary Incontinence; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: Perineal-applied electrical stimulation shaped for males.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment group (Experimental): Self-applied electrical stimulation for 6 weeks.
  Interventions: Device: Perineal-applied electrical stimulation

INTERVENTIONS:
Device: Perineal-applied electrical stimulation — Small controller that outputs stimulation for stress incontinence and OAB, attached to a male-anatomy thin GelPad placed in the perineal area.
  Other Names: Elidah; Elitone; Edytone

SUMMARY:
The purpose of this research is to evaluate the effectiveness of the Elidah neuromuscular stimulation treatment to reduce incontinence in men post-prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for robotic-assisted laparoscopic prostatectomy
* Read and speak English
* Predominant SUI of at least 1 pad/day

Exclusion Criteria:

* History or symptoms of urinary incontinence, urinary retention, extra-urethral incontinence, overflow incontinence
* Complete denervation of the pelvic floor
* Severe Obesity as defined by BMI >= 40
* Has undergone pre-op pelvic floor exercise strengthening
* Pelvic pain/painful bladder syndrome
* Implanted cardiac device, untreated cardiac arrhythmia or suffer from other heart problems.
* History of epilepsy
* Underlying neurologic/neuromuscular disorder
* Metal implants in the abdomen or pelvic area
* Chronic coughing
* Impaired decision making, suicidal thoughts, or drug/alcohol dependence
* Uncontrolled intercurrent illness that would limit compliance with study requirements
* Lacks capacity to adhere with study requirements
* Lacks capacity to consent for themselves.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Leakage by Pad weight | 6 weeks
  24-hr pad weight

SECONDARY OUTCOMES:
Safety measured by no Adverse events | 6 weeks
  No adverse events
Quality of Life Improvement | 6 weeks
  Incontinence I-QoL survey
Quality of Life Improvement | 6 weeks
  Sexual Health SHIM survey
Reduction in leakage | 6 weeks
  As measured by Pads per day
Reduction in leakage at Night | 6 weeks
  As measured by Nocturia episode
Reduction in leakage | 6 weeks
  As measured by daytime leaking episodes

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Kolb, MS,MBA, Principal Investigator — Elidah, Inc.
Locations (1):
- Elidah, Monroe, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided